CLINICAL TRIAL: NCT06115278
Title: Pain Rating Challenges and Patterns
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Erin Dannecker, Associate Professor & Director Of Scholarly Activity, University of Missouri-Columbia
Other Study IDs: 2091563
Record Dates: First submitted 2023-10-25; First posted 2023-11-02 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- nurses: Our inclusion criteria for the nurses are the following: (1) 18 years old or older; (2) currently employed as a licensed nurse; and (3) current employment duties include routinely assessing the musculoskeletal pain of cognitively intact, adult outpatients. Our exclusion criteria for the nurses are the following: (1) currently managing a painful musculoskeletal condition; and (2) has ever felt musculoskeletal pain on most days for 3 months or longer.
  Interventions: Other: survey
- patients: Our inclusion criteria for the patients are the following: (1) 18 years old or older; (2) currently being treated by a health care provider for a painful musculoskeletal condition; (3) has felt a usual musculoskeletal pain intensity rating of "2" or higher on a "0" to "10" scale over the last 24 hours; (4) has felt extreme pain that completely disappeared; (5) has felt musculoskeletal pain on most days of the last 3 months; (6) chronic musculoskeletal pain has increased and decreased during the last 3 months; and (6) has felt musculoskeletal pain in more than one location on most days of the last 3 months. Our exclusion criterion for the patients is ever employed as a licensed health care provider.
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — survey

SUMMARY:
Our long-term goal is to improve pain communication for patients' health. For this project, we seek information on patients' and health care nurses' (1) mental effort when choosing or understanding, respectively, pain intensity ratings, and (2) confidence in the accuracy of pain intensity rating patterns. This information will clarify the importance of mental effort from pain ratings and the probability of pain intensity rating patterns.

Our primary aim will compare patients' and nurses' perceptions of the mental effort of choosing (Aim 2a) and understanding (Aim 2b) pain intensity ratings. We hypothesize that patients will rate mental effort higher than nurses for choosing ratings and lower than nurses for understanding ratings. The results will inform future efforts to improve pain communication between patients and nurses.

DETAILED DESCRIPTION:
Our long-term goal is to improve pain communication for patients' health. For this project, we seek information on patients' and health care nurses' {1} mental effort when choosing or understanding, respectively, pain intensity ratings, and {2} confidence in the accuracy of pain intensity rating patterns. This information will clarify the importance of mental effort from pain ratings and the probability of pain intensity rating patterns.

Aim 1 {exploratory} will compare the mental effort of choosing {Aim 1a} and understanding {Aim1b different pain intensity rating scales. We hypothesize mental effort will be lower for {a} the "worst pain you have ever felt" scale than "worst pain you can think of" scale, {b} a 7-day recall period than a 1-month recall period, and {c} focus on one body area than summarizing across body areas. The results will clarify the impact of pain intensity scales' characteristics on mental effort.

Aim 2 {primary} will compare patients' and nurses' perceptions of the mental effort of choosing {Aim 2a} and understanding {Aim 2b} pain intensity ratings. We hypothesize that patients will rate mental effort higher than nurses for choosing ratings and lower than nurses for understanding ratings. The results will inform future efforts to improve pain communication between patients and nurses.

Aim 3 {exploratory} will determine the relationship between perceptions of mental effort and the importance of decreasing that mental effort for patients {Aim 3a} and nurses {Aim 3b}. We hypothesize perceptions of mental effort will positively correlate with the importance of decreasing mental effort. The results will clarify the importance of mental effort for pain intensity ratings.

Aim 4 {exploratory} will evaluate the equivalence of patients' and nurses' confidence in the accuracy of fictional pain intensity rating patterns. We hypothesize that patients' and nurses' confidence in the accuracy will be equally low because the patterns tested should be improbable. Future studies may investigate the ability of improbable pain intensity rating patterns to evaluate the usability and psychometrics of pain measures.

Aim 5 {exploratory} will test the relationship between confidence in the accuracy of fictional pain intensity rating patterns and the importance of increasing that confidence for patients {Aim 5a} and nurses {Aim 5b}. We hypothesize confidence will negatively correlate with the importance of increasing confidence. The results will clarify the importance of confidence in pain intensity rating accuracy.

ELIGIBILITY:
Our inclusion criteria for the patients are the following:

* 18 years old or older;
* currently being treated by a health care provider for a painful musculoskeletal condition;
* has felt a usual musculoskeletal pain intensity rating of "2" or higher on a "0" to "10" scale over the last 24 hours;
* has felt extreme pain that completely disappeared;
* has felt musculoskeletal pain on most days of the last 3 months;
* chronic musculoskeletal pain has increased and decreased during the last 3 months; and
* has felt musculoskeletal pain in more than one location on most days of the last 3 months.

Our exclusion criterion for the patients is:

• ever employed as a licensed health care provider.

Our inclusion criteria for the nurses are the following:

* 18 years old or older;
* currently employed as a licensed nurse; and
* current employment duties include routinely assessing the musculoskeletal pain of cognitively intact, adult outpatients.

Our exclusion criteria for the nurses are the following:

* currently managing a painful musculoskeletal condition; and
* has ever felt musculoskeletal pain on most days for 3 months or longer.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic pain & nurses without chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-02-24 (Actual); Study Completion 2024-02-24 (Actual)

PRIMARY OUTCOMES:
mental effort | baseline
  ordinal self-report of expected amount of thought allocated to choosing a numeric pain intensity rating; higher scores mean more mental effort
importance of decreasing mental effort | baseline
  ordinal self-report of importance of decreasing amount of thought allocated to choosing or understanding a numeric pain intensity rating; higher scores mean more importance

SECONDARY OUTCOMES:
confidence in the accuracy of fictional pain intensity ratings | baseline
  ordinal self-report of confidence in numeric pain intensity ratings; higher scores mean more confidence

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri - Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided